CLINICAL TRIAL: NCT03574155
Title: Impact of Preoperative Counseling and Education in Reducing Anxiety Levels in Patients With Gynecologic Tumors: A Prospective Randomized Study
Brief Title: Impact of Preoperative Counseling and Education in Reducing Anxiety Levels in Patients With Gynecologic Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ricardo dos Reis, Principal investigator, Barretos Cancer Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 81886517000005437
Record Dates: First submitted 2018-06-05; First posted 2018-06-29 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Anxiety Disorders
Keywords: Gynecological cancer; Anxiety; Pre-operative counseling
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Intervention Model Description: Group control Pre-operative Orientation Routine Application of the questionnaire (ESAS) and (HADS)
  Experimental Group Pre-operative Counseling and Education Application of the questionnaire (ESAS) and (HADS)
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control- group (No Intervention): It is composed of patients scheduled for surgical treatment by tumors of the uterine cervix, vulva, ovary or endometrium, who will receive preoperative and postoperative guidelines according to the usual routine for the perioperative period of the present institution. Patients and their followers of the control group will participate in a preoperative consultation with the surgeon to discuss the indication of the procedure and its risks, benefits and alternatives to the procedure being indicated, if any.
  Pre-operative Counseling and Education Application of the questionnaire (ESAS) and (HADS)
- Experimental Group (Experimental): Composed of patients scheduled for surgical treatment by tumors of the uterine cervix, vulva, ovary or endometrium who will receive preoperative counseling and education through a pre-defined protocol after preoperative consultation with the surgeon. The counseling session will take place with at least one companion. The purpose of this session is to supplement, re-emphasize and strengthen the perioperative guidelines. An illustration (explanatory folder) will be used to demonstrate the location of the surgery, how the scar will be and on which sites of the abdomen and organs the surgery will cover. All this counseling and education will be applied at the same time to the patient and her companion. At the end of the intervention, a space will be left open for both the patient and the companion to ask questions and questions.
  Pre-operative Counseling and Education Application of the questionnaire (ESAS) and (HADS)
  Interventions: Behavioral: Pre-operative Counseling and Education

INTERVENTIONS:
Behavioral: Pre-operative Counseling and Education — Group control Pre-operative Orientation Routine Application of the questionnaire (ESAS) and (HADS) Post-operative Immediate (1 OP) Application of the Questionnaire to assess HADS and ESAS Anxiety (Patient)
  Experimental Group Pre-operative Counseling and Education Application of the questionnaire (ESAS) and (HADS)
  Late postoperative (2 - 4 weeks) Questioning the patient and companion evaluating the degree of satisfaction regarding the preoperative guidelines.
  Other Names: Application of the questionnaire (ESAS) and (HADS)
  Arms: Experimental Group

SUMMARY:
The surgical procedure can be considered a transition in the patient's life. The transition can generate instability and produce negative effects, which may be temporary or permanent. Failure to prepare people to deal with the unexpected, such as diagnosing a disease, such as cancer, and surgical necessity can be a frightening and frustrating experience, developing painful and distressing feelings, involving their family members as well.

DETAILED DESCRIPTION:
A preoperative orientation process with potential benefits to the patient has been adopted for some surgical procedures. However, recently some surgical specialties such as orthopedics have been implemented in their routine a potentially modifiable conduct of the emotional trauma of a surgery, is the use of the preoperative advice and orientation, in order to attain an ability to increase the client's satisfaction, to facilitate the recovery, decrease the rate of complications without increasing reintegration, decrease hospitalization time and health costs without additional patient risk. There is a belief among surgeons that preoperative counseling and counseling is vitally important for a post-operative outcome. Despite this, there is a paucity of well-conducted studies that examine the importance of the need for preoperative counseling with detailed information to analyze the yearnings and needs as well as the emotional impact. In addition, there are few studies evaluating the emotional impact and impact in the postoperative period in general of detailed preoperative counseling in patients with gynecological tumors submitted to laparotomy and minimally invasive surgery. For these reasons, this study aims to evaluate whether the application of detailed and clear preoperative counseling and education about the surgical procedure to be performed, as well as all the perioperative guidelines that involve the procedure versus the usual preoperative orientation and preoperative, can have an impact on the level of anxiety of the patient and the companion, as well as assess the degree of satisfaction of the companion.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to accessory treatment for tumors of the cervix, vulva, ovary or endometrium.
* Primary therapy, which may be radiotherapy or chemotherapy.
* Patients between the ages of 20 and 80 years.
* Patients submitted to a laparotomic or minimally invasive method (robotic and laparoscopic).
* Patients should be treated at the Oncology Gynecology Service of the Barretos Cancer Hospital.

Exclusion Criteria:

* Patients treated at another oncology service previously.
* Patients who have already been treated for some other cancer in the past.
* Patients without a complete primary level and / or who can not read or write.
* Patients and / or family members who refuse to participate in the study.
* Patients who will be admitted to the ICU.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | up to 2 months
  The investigators will measure anxiety levels using the Hospital Anxiety and Depression Scale.The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal.

CONTACTS AND LOCATIONS:
Locations (1):
- Ricardo Reis, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No